CLINICAL TRIAL: NCT05632887
Title: The Effect of Eyeliner on Tear Composition, Tear Secretion and Tear Film Stability：a Prospective Cohort Study.
Brief Title: The Effect of Eyeliner on Tear Composition, Tear Secretion and Tear Film Stability.
Status: Recruiting | Type: Observational
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20220920E
Record Dates: First submitted 2022-10-09; First posted 2022-12-01 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — tears
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control: The population who do not use eyeliner.
  Interventions: Other: no intervention
- Eyeliner: The population who using eyeliner and the duration and frequency are appropriate。
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Eyeliner is one of the most common eye cosmetics. The main ingredients are titanium oxide, pigment, grease and preservative. The user will apply the eyeliner to the eyelid and eyelash. With the blinking again and again, the components of the eyeliner may enter the tear film and continue to act on the eye surface. Therefore, the investigators suspect that the use of eyeliner may be an important factor leading to dry eye disease. In order to explore the relationship between the use of eyeliner and dry eye disease, the investigators plan to collect eye surface characteristic data of the two groups of people who use eyeliner and who do not use it.Then use Raman analysis to explore whether the use of eyeliner will lead to changes in tear composition.The investigators intend to analyze the difference of tear composition between the two groups to understand the relationship between the change of tear composition and tear film stability.So that the investigators can identify the risk factors of dry eye disease, and provide basis for prevention and early treatment.

DETAILED DESCRIPTION:
The investigators will include the population according to the inclusion criteria and exclusion criteria.The subjects in the eyeliner group and the control group filled in the survey to score the ocular surface disease index. Tear secretion test and sodium fluorescein staining are conducted in the eyeliner group and the control group, and the results are recorded. The intraocular pressure of the two groups is measured and recorded. Dry eye analysis is conducted for the two groups of people to collect relevant data. Tears are collected by capillary glass tube and stored for further Raman analysis.

ELIGIBILITY:
Inclusion Criteria:

* People aged 20-35 who use eyeliner or do not use eyeliner .
* People who use eyeliner have used it for ≥ 1 year; Frequency ≥ 3 times/week.

Exclusion Criteria:

* Other serious systemic diseases.
* Other systemic diseases related to ocular surface, such as rheumatoid arthritis, systemic lupus erythematosus, Sjogren's syndrome and other immune system diseases or other eye diseases, history of eye surgery and trauma.
* Lactating women or pregnant women.
* Use electronic products for more than 4 hours every day.
* Patients with circadian rhythm disorder.
* People with radiation exposure history.
* Non permanent residents in Wuhan.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The main population of our study is the young women who do not have other diseases that affect the health of eye surface and use or do not use eyeliner.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2022-11-20 (Actual); Primary Completion 2026-09-15 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
The Schirmer's test evaluates aqueous tear production. | baseline
  Schirmer test is a simple method to measure the amount of tear secretion.It is helpful in the assessment of patients with signs and/or symptoms of dry eye as it can determine whether surface dryness is due to reduced tear production from the lacrimal glands as opposed to some other cause.Normal aqueous tear production is supported by measurements of > 15 mm after 5 minutes.Mild-moderate reduction of aqueous production: 5mm-14mm after 5 minutes.Severe dryness due to reduced tear production is <5mm after 5 minutes.
The gland loss assessed by meibography images. | baseline
  The investigators can observe the morphology of meibomian gland to grade the degree of Dry Eye.The morphology was evaluated by analyzing meibography images obtained with the non-contact infrared meibography system OCULUS Keratograph 5.MG loss in each eyelid was evaluated subjectively using a four-point grading scale (meibograde) of 0-3described as : grade 0: 0-25% loss; grade 1: 26-50% loss; grade 2: 51-75% loss; and grade 3: >75% loss.
Evaluation of lipid content and ionic composition in tears by raman analysis. | baseline
  The investigators can use Raman spectroscopy to compare the changes of tear composition between the two groups.Raman spectroscopy is a technique that detects vibrational motions in molecules and can be used for lipids. It is a powerful technique and often used when analyzing biological samples such as lipids and proteins because it's non-invasive, highly accurate, insignificant amount and provides abundant chemical information.The fatty acids, triglycerides, phospholipids, sphingolipids, cholesterol and carotenoids can be detected.And the investigators can use a special instruments to test Na+,K+,Mg2+ and Cl- those are very important in tear film homeostasis.

CONTACTS AND LOCATIONS:
Overall Officials: Min Ke, Study Chair — Ophthalmology Department of Zhongnan Hospital of Wuhan University
Locations (1):
- Zhongnan Hospital of Wuhan University, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No